CLINICAL TRIAL: NCT01018251
Title: Monitoring Treatment Response in Women With Breast Cancer Utilizing FLT-PET/CT
Brief Title: Positron Emission Tomography in Monitoring Treatment Response in Women With Newly Diagnosed Breast Cancer
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Sponsor: Abramson Cancer Center at Penn Medicine (Other)
Responsible Party: Julia Tchou, MD, Abramson Cancer Center of the University of Pennsylvania
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: UPCC 01109
Record Dates: First submitted 2009-11-18; First posted 2009-11-23 (Estimated); Last update posted 2015-12-15 (Estimated); Status verified 2015-12

CONDITIONS: Adult Women With a New Diagnosis of Invasive Breast Cancer (Have Not Undergone Treatment)
MeSH Terms: interventions — alovudine; Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Arm I (Experimental): Patients undergoing definitive surgery after cancer diagnosis undergo 3'-deoxy-3'-[18F] fluorothymidine (FLT)-PET prior to definitive surgery. Patients undergoing neoadjuvant chemotherapy prior to definitive surgery undergo FLT-PET prior to and after completion of neoadjuvant chemotherapy
  Interventions: Other: 3'-deoxy-3'-[18F]fluorothymidine; Procedure: Positron Emission Tomography/computed tomography; Radiation: FLT-PET/CT

INTERVENTIONS:
Other: 3'-deoxy-3'-[18F]fluorothymidine — Given IV
  Other Names: 18F-FLT
Procedure: Positron Emission Tomography/computed tomography
Radiation: FLT-PET/CT

SUMMARY:
This study will investigate the sensitivity and specificity of FLT-PET/CT in primary breast cancer detection and in the use of FLT-PET in monitoring how well a breast tumor respond to treatment. We will compare this technique with other imaging modalities as well as with tissue collection (during a biopsy). We will recruit women with a newly diagnosed invasive breast cancer, who are able to tolerate undergoing a PET/CT (possibly two scans) scan,

DETAILED DESCRIPTION:
Our overall goal is to use this clinical trial as a platform to validate fibroblast activation protein (FAP) as a biomarker for the tumor microenvironment and to explore the dynamic interaction between proliferating tumor cells and the tumor microenvironment. Our long term goal is to develop new drugs that will target the tumor microenvironment as novel therapeutic and chemoprevention strategies.

ELIGIBILITY:
Inclusion Criteria:

* Breast biopsy positive for an invasive malignancy (core needle, mammatone, or incisional biopsy)
* Participants must be planning to have surgery at the Hospital of the University of Pennsylvania
* Participants must be able to tolerating lying on the table for about an hour
* Newly diagnosed primary breast cancer, which is classified as being operable (T1-T4)

Exclusion Criteria:

* Pregnant women
* History of severe renal disease
* Prior history of breast cancer of the study breast within the last five years.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2009-03; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Sensitivity and specificity of FLT-PET comparing with standard FDG-PET
Correlate SUV with % Ki67 nuclear stain

SECONDARY OUTCOMES:
Change in SUV with change in tumor proliferation index (%Ki67 nuclear stain) (when neoadjuvant therapy is used)
Tumor volume pre and post chemotherapy as assessed by clinical exam, breast imaging studies, histopathological examination, and breast cancer outcome parameters (when neoadjuvant therapy is used)